CLINICAL TRIAL: NCT01946724
Title: PERSPECTIVE: Percutaneous Revascularization at Piedmont for Chronic Total Occlusions Survey
Brief Title: In-hospital and Long-term Outcomes for Percutaneous Chronic Total Coronary Occlusion Revascularization in a High-volume, Multi-operator Program
Acronym: Perspective
Status: Completed | Type: Observational
Sponsor: Piedmont Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: Perspective
Record Dates: First submitted 2013-09-12; First posted 2013-09-20 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study whether percutaneous chronic total occlusion (CTO) revascularization, by the use of Percutaneous Coronary Intervention (PCI), stenting, guidewire, and catheter, improves a patient's quality of life and their left ventricular function, reduces angina severity, and improves long-term survival.

DETAILED DESCRIPTION:
The purpose of this study is to study whether percutaneous chronic total occlusion (CTO) revascularization, by the use of Percutaneous Coronary Intervention (PCI), stenting, guidewire, and catheter, improves a patient's quality of life and their left ventricular function, reduces angina severity, and improves long-term survival. The study will consist of the two following groups:

Retrospective patients This group will consist of consecutive patients that have already undergone CTO PCI by the PHI CTO team.

* The patients will be contacted by telephone for informed consent and will be asked how they are feeling and if they have seen any doctors for their heart conditions. The patient will also be asked if they are taking antiplatelet medicines as prescribed, and if there have been any changes in on their medicines.
* If more than 12 months have passed since the procedure, the patients will be queried regarding medical history
* If the patient cannot be contacted, then analysis of data will be limited to de-identified data collected from the chart, procedure angiogram, and the procedure report.

Prospective patients This group will consist of patients in which the CTO procedure will be performed by the PHI CTO team.

* A clinical assessment will be performed before the stent procedure
* A blood sample will be taken for routine blood chemistry and hematology
* Medications will be prescribed to prevent blood clots
* Follow-up will occur 6 and 12 months post-procedure

ELIGIBILITY:
Inclusion Criteria:

1. The subject is > 18 years of age at the time of consent
2. Subjects experiencing clinical symptoms considered suggestive of ischemic heart disease (eg, chest pain or discomfort or symptoms considered by the investigator to represent anginal equivalents) or having evidence of myocardial ischemia (eg, abnormal functional study) attributed to the CTO target vessel and scheduled for clinically indicated percutaneous CTO revascularization or are subjects with multi-vessel disease and/or Acute Coronary Syndrome (ACS) that are undergoing a staged CTO PCI procedure with the intent to achieve complete revascularization.
3. Subject must have at least 1 target segment meeting non-acute total coronary occlusion as defined below. A CTO is any non-acute total coronary occlusion fulfilling the following angiographic characteristics and:

   1. High-grade native coronary stenosis
   2. Thrombolysis in Myocardial Infarction (TIMI) 0 or 1 antegrade flow
   3. Estimated in duration at least 3 months by clinical history and/or comparison with antecedent angiogram, functional study or electrocardiogram
   4. CTO segment may be de novo or previously treated via PCI
4. Subject is eligible and consents to undergo or has undergone a PCI procedure
5. Subject is an acceptable candidate for percutaneous transluminal coronary angioplasty (PTCA) and stenting.
6. Subject is willing and able to provide informed consent as approved by local Institutional Review Board/Ethics Committee and to complete the protocol requirements for the study.
7. Female subjects of child-bearing potential with a negative qualitative or quantitative pregnancy test in accordance to the Piedmont Hospital Policy.

Exclusion Criteria:

1. Any known allergy, hypersensitivity or contraindication to iodinated contrast that cannot be effectively managed medically
2. Any known allergy, hypersensitivity or contraindication to clopidogrel bisulfate (Plavix®), prasugrel (Effient®) or ticagrelor (Brilinta®)-- for which alternative agents cannot be used-- or aspirin, heparin, nickel, stainless steel, zotarolimus, or everolimus
3. Any contraindication to cardiac catheterization or to any of the standard concomitant therapies used during routine cardiac catheterization and PCI
4. Subjects with any other pathology or indication which in the opinion of the investigator, might put the subject at risk, preclude follow-up, or in any way confound the results of the study
5. Known previous medical condition yielding expected survival less than one year
6. Subjects who are unable or unwilling to comply with the protocol or not expected to complete the study period, including its follow-up requirements
7. Subjects with evidence of ongoing or active clinical instability including any of the following:

   1. Sustained systolic blood pressure < 100 mmHg (if different from baseline) or cardiogenic shock
   2. Acute pulmonary edema that has not been medically stabilized
   3. Suspected acute myocarditis, pericarditis, endocarditis, or cardiac tamponade
   4. Suspected dissecting aortic aneurysm
8. Subjects with known clinically significant abnormal laboratory findings including:

   1. White Blood Cells (<1,000 WBC/mm3)
   2. Thrombocytopenia (<100,000 platelets/mm3)
9. Subjects with history of bleeding diathesis or coagulapathy or refusal of blood transfusions
10. Female subjects of child-bearing potential with a positive qualitative or quantitative pregnancy test or with a negative qualitative or quantitative pregnancy test who plan to become pregnant within 12 months of enrolling in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects experiencing clinical symptoms considered suggestive of ischemic heart disease or having evidence of myocardial ischemia who have had or are scheduled to have percutaneous chronic total occlusion (CTO) revasulcarization by Percutaneous Coronary Intervention (PCI)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
CTO procedural success | 1 year
  CTO procedural success as defined by an achievement of a final residual angiographic stenosis < 50% within the treated segment with >=TIMI 2 antegrade flow.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events (MACE) | Prior to Index Hospitalization Discharge (< 1 year from procedure)
  The occurrence of major adverse cardiac events (MACE): death, myocardial infarction, and repeat target lesion revascularization (TLR) prior to index hospitalization discharge (< 1 year from procedure)
Clinical Outcomes | 1 year
  Compare 1-year clinical outcomes among patients treated with zotarolimus-eluting stents with a performance goal derived from prior chronic total occlusion drug-eluting stent trials

OTHER OUTCOMES:
MACE | 1 year
  1-year composite clinical outcome of MACE among all subjects undergoing attempted CTO revascularization that are enrolled in the study.

CONTACTS AND LOCATIONS:
Overall Officials: David Kandzari, MD, Principal Investigator — Piedmont Heart Institute
Locations (1):
- Piedmont Heart Institute, Atlanta, Georgia, United States